CLINICAL TRIAL: NCT00587340
Title: A Survey of Sleep Problems in Survivors of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York Presbyterian Hospital (Other); Rockefeller University (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 06-071
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 15 subjects with subjective sleep disturbance based on the Pittsburgh Sleep Quality Index
- 2: mild/moderate subjective sleep disturbance (insomnia) based on the Pittsburgh Sleep Quality Index
- 3: severe subjective sleep disturbance (insomnia)based on the Pittsburgh Sleep Quality Index

SUMMARY:
The purpose of this study is to gain greater understanding of the problems breast cancer survivors experience related to difficulty sleeping and insomnia. Poor sleep can affect a person's mood, increase feelings of fatigue, as well as pain. A greater knowledge and understanding of sleep disturbances can lead to more effective treatment of sleep problems and significantly improve quality of life.

DETAILED DESCRIPTION:
Individuals who consent to participate in this study will be asked to complete a battery of questionnaires that will take approximately 1 hour. Based on answers they give to the questionnaires, 45 patients will be asked to participate in a sleep study done at a sleep lab.

If you choose to take part, then you will be asked to do the following:

Spend approximately 1 hour answering questionnaires either at the breast cancer center with a research assistant, at home on the phone with a research assistant, or by completing the questionnaires at home and returning them by mail. You will only be asked to complete questionnaires one time. The questionnaires will ask you questions about your:

* Past medical history
* Demographics
* Sleep quality
* Sleep habits
* Energy level, pain, daytime sedation
* Quality of life
* Menopausal symptoms
* Depression
* Fears

If you are then selected to participate in the sleep study, further information will be provided for you.

After you are finished with the questionnaires, the research assistant will provide you with any necessary further information and feedback. The research assistant will also be able to put you in contact with a study doctor should you require any further assistance. After you are finished with the study, the study doctor may contact you for clarification of your answer on a question, or for an answer if you have by any chance missed a question.

ELIGIBILITY:
Inclusion Criteria:

Subject Inclusion Criteria for Questionnaire Portion of Study

* Women with a diagnosis of Stage I, II, or III breast cancer who are one year posttreatment, but not more than 10 years post-treatment (surgery, chemotherapy, and/or radiation) prior to entrance into the study. Use of biological and/or hormonal therapy is acceptable.
* Greater than 18 years of age.
* Able to speak and read English.

Exclusion Criteria:

Subject Exclusion Criteria for Questionnaire Portion of Study •Evidence of acute or chronic encephalopathy or psychiatric disease severe enough to compromise data collection.

Exclusion Criteria for Sleep Lab Study

•Women who are unable or unwilling to avoid alcohol, caffeine consumption or cigarette smoking as of 3 p.m. on the day of the sleep study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2006-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of cancer-related insomnia in women surviving breast cancer (Stage I, II, & III) who are at least one year, but not more than 10 years posttreatment & to study its deleterious impact on qol | 2 years
To describe the underlying physiology and nature of sleep disturbances in this cohort of women by performing sleep lab studies with a subset of the sample | 2 years

SECONDARY OUTCOMES:
To survey the medical, demographic and psychosocial correlates of cancer-related insomnia in this cohort of women to identify subgroups with potentially differing etiologies and associated symptoms to help plan relevant intervention studies | 2 Years
To preliminarily describe correlations between subgroups and sleep disturbances documented in the sleep lab studies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Passik, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org